CLINICAL TRIAL: NCT01463397
Title: Multinational, Multicenter, Randomized Double-Blind, Placebo-Controlled, Parallel-Group Study of Efficacy and Safety of SAR292833 Administration for 4 Weeks in Patients With Chronic Peripheral Neuropathic Pain
Brief Title: Efficacy and Safety of SAR292833 Administration for 4 Weeks in Patients With Chronic Peripheral Neuropathic Pain
Acronym: Alchemilla
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT11917; 2011-001876-21 (EudraCT Number); U1111-1120-0404 (Other: UTN)
Record Dates: First submitted 2011-10-28; First posted 2011-11-01 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SAR292833 dose level 1 (Experimental): Dose level 1 twice daily immediately after breakfast/dinner
  Interventions: Drug: SAR292833
- SAR292833 dose level 2 (Experimental): Dose level 2 twice daily immediately after breakfast/dinner
  Interventions: Drug: SAR292833
- Placebo (Placebo Comparator): Placebo (for SAR292833) twice daily immediately after breakfast/dinner
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SAR292833 — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: SAR292833 dose level 1; SAR292833 dose level 2
Drug: placebo — Pharmaceutical form:capsule
  Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objective:

To assess the efficacy of SAR292833 versus placebo in reducing pain intensity associated with chronic peripheral neuropathic pain using 11-point numerical rating scale (NRS).

Secondary Objectives:

* To compare the effects of SAR292833 with placebo on the change of neuropathic pain symptoms versus baseline Neuropathic Pain Symptoms Inventory (NPSI);
* To evaluate the effects of SAR292833 in comparison to placebo on the change in pain intensity of mechanical allodynia;
* To investigate the safety and tolerability of SAR292833 in comparison to placebo;
* To investigate the pharmacokinetics (PK) and the relationships between main efficacy parameters or pharmacodynamic effect (PD) and pharmacokinetics (PK/PD) of SAR292833 in patients with chronic peripheral neuropathic pain.

DETAILED DESCRIPTION:
Total study duration (from screening to last follow-up visit) is 9 weeks that includes a 3 week follow-up period.

ELIGIBILITY:
Inclusion criteria:

-The study will include adult patients of either gender, 18 - 85 of age, who have signed the informed consent form, and presenting with chronic peripheral neuropathic pain associated with: diabetic polyneuropathy, post-herpetic neuralgia.

* The neuropathic pain must have a distinct neuroanatomically plausible distribution with sensory signs and symptoms confirmed by DN4 (Douleur Neuropathique en 4 questions) score of ≥4 and being present for more than 3 months.
* SAR292833 should be taken in fed condition. Therefore, only patients who were judged to be reliable to fulfill this condition (used to having breakfast and dinner) will be included in the study.

Exclusion criteria:

* Patients with a baseline average daily pain intensity for their neuropathic pain < 5 on the 11-point NRS over the last 7 days before randomization;
* Patients with a pain intensity of ≥ 9 on the 11-point NRS at Visit 1;
* Any pain other than the neuropathic pain of equal or greater severity;
* Sensory polyneuropathy post chemotherapy or in the context of cancer or AIDS;
* Patients with complex regional pain syndrome;
* Trigeminal neuralgia;
* Patients with clinically significant or uncontrolled hepatic, metabolic, gastrointestinal, cardiovascular, respiratory, neurological (other than neuropathy), psychiatric, hematological, renal, or dermatological disease, or any other medical condition that might interfere with the evaluation of study medication according to Investigator's medical judgment;
* Patients on statins metabolized by CYP3A4, (e.g. simvastatin, atorvastatin) and abnormal CPK level;
* Major depression;
* Serum creatinine >150 μmol/L;
* ALT 3 x ULN;
* Total bilirubin > 1.5 x ULN except known Gilbert syndrome;
* Presence of signs of clinically significant abnormalities on a standard electrocardiogram (ECG) recording at the screening visit according to Investigator's medical judgment;
* Pregnant or breastfeeding women;
* Women of childbearing potential (WOCBP), not protected by highly effective contraceptive method of birth control;
* Patients with diabetes mellitus and time between diagnosis of diabetes and enrolment <6 months;
* Patients with diabetes mellitus and HbA1c >10% or fasting plasma glucose >250 mg/dL;
* Use of the following drugs within 7 days prior to start with the pain intensity assessment (Visit 2):
* Antidepressants (except for stable [>30 days] regimens of Selective serotonin reuptake inhibitors (SSRIs) for treatment of anxiety or depression), anticonvulsants or mexiletine for the treatment of pain;
* Opioids or morphinomimetics;
* Fatty acid supplements, primrose oil, myoinositol, chromium picolinate that are known to be used in neuropathic pain;
* Acetyl salicylic acid (ASA) except up to 325 mg/d for myocardial infarction or transient ischemic attack prophylaxis;
* Benzodiazepines other than indicated at low doses for sleep disorders;
* Capsaicin patch;
* Lidocaine patch;
* Electroconvulsive therapy within 30 days of baseline evaluation;
* CYP3A4 potent and moderate inhibitors;
* CYP3A4 potent and moderate inducers;
* Substrates of CYP3A4 with narrow therapeutic window.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average daily pain intensity as measured by the 11-point NRS; | Baseline to 4 weeks
  The average daily pain intensity is the mean of the last consecutive 7 days.

SECONDARY OUTCOMES:
Percentage of patients with reduction in pain intensity of at least 30% and 50% at endpoint compared to baseline derived from the primary efficacy endpoint; | Baseline to 4 weeks
Change in Neuropathic Pain Symptom Inventory (NPSI) after 4 weeks treatment compared to baseline | Baseline to 4 weeks
Change in intensity of the mechanical allodynia after 4 weeks treatment compared to baseline using visual analog scale (VAS) | Baseline to 4 weeks
Amount of and time to first rescue medication intake during the treatment period. | 4 weeks
Change in Daily Sleep Interference Score (DSIS), clinical global impression of change (PGIC and CGIC). | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (61):
- United States (28):
  - Investigational Site Number 840014, Tucson, Arizona
  - Investigational Site Number 840007, Garden Grove, California
  - Investigational Site Number 840020, Newport Beach, California
  - Investigational Site Number 840038, Santa Ana, California
  - Investigational Site Number 840002, Tustin, California
  - Investigational Site Number 840046, Coral Gables, Florida
  - Investigational Site Number 840013, Ocala, Florida
  - Investigational Site Number 840034, Palm Beach Gardens, Florida
  - Investigational Site Number 840019, Evansville, Indiana
  - Investigational Site Number 840012, Indianapolis, Indiana
  - Investigational Site Number 840042, Framingham, Massachusetts
  - Investigational Site Number 840004, Springfield, Massachusetts
  - Investigational Site Number 840035, St Louis, Missouri
  - Investigational Site Number 840010, Las Vegas, Nevada
  - Investigational Site Number 840037, Albuquerque, New Mexico
  - Investigational Site Number 840040, Hartsdale, New York
  - Investigational Site Number 840001, New York, New York
  - Investigational Site Number 840033, Rochester, New York
  - Investigational Site Number 840015, Raleigh, North Carolina
  - Investigational Site Number 840022, Winston-Salem, North Carolina
  - Investigational Site Number 840017, Toledo, Ohio
  - Investigational Site Number 840044, Altoona, Pennsylvania
  - Investigational Site Number 840018, Johnstown, Pennsylvania
  - Investigational Site Number 840045, Tullahoma, Tennessee
  - Investigational Site Number 840006, Austin, Texas
  - Investigational Site Number 840043, Dallas, Texas
  - Investigational Site Number 840032, Dallas, Texas
  - Investigational Site Number 840016, Seattle, Washington
- Czechia (3):
  - Investigational Site Number 203002, Olomouc
  - Investigational Site Number 203005, Prague
  - Investigational Site Number 203006, Prague
- Hungary (6):
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348005, Budapest
  - Investigational Site Number 348007, Budapest
  - Investigational Site Number 348002, Budapest
  - Investigational Site Number 348006, Debrecen
  - Investigational Site Number 348003, Zalaegerszeg
- Poland (4):
  - Investigational Site Number 616001, Bydgoszcz
  - Investigational Site Number 616002, Lublin
  - Investigational Site Number 616007, Sandomierz
  - Investigational Site Number 616004, Włocławek
- Russia (13):
  - Investigational Site Number 643006, Kazan'
  - Investigational Site Number 643007, Kazan'
  - Investigational Site Number 643008, Moscow
  - Investigational Site Number 643010, Moscow
  - Investigational Site Number 643009, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643011, Moscow
  - Investigational Site Number 643004, Nizhny Novgorod
  - Investigational Site Number 643012, Novosibirsk
  - Investigational Site Number 643013, Saint Petersburg
  - Investigational Site Number 643003, Saint Petersburg
  - Investigational Site Number 643014, Saint Petersburg
  - Investigational Site Number 643005, Yaroslavl
- Slovakia (3):
  - Investigational Site Number 703004, Banská Bystrica
  - Investigational Site Number 703001, Dubnica nad Váhom
  - Investigational Site Number 703003, Krompachy
- Ukraine (4):
  - Investigational Site Number 804002, Kiev
  - Investigational Site Number 804005, Kiev
  - Investigational Site Number 804004, Kyiv
  - Investigational Site Number 804003, Kyiv